CLINICAL TRIAL: NCT05029674
Title: Use of Biometric Data to Understand Surgeon Performance, Strain, and Recovery
Brief Title: Understanding Performance: Enhancing Recovery as Surgeons
Acronym: ERAS
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Cindy Kin, Assistant Professor of Surgery, Stanford University
Other Study IDs: 58625
Record Dates: First submitted 2021-08-17; First posted 2021-08-31 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Burnout, Professional
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Whoop — Wear WHOOP Strap, complete surveys

SUMMARY:
Reliably achieving peak performance requires balancing the strain of the prior day with sufficient recovery to be ready for the next day. Surgery has a long standing tradition long hours of hard work often at the expense of adequate sleep. Decreased sleep and recovery has physiologic consequences which can be measured using biometric data. The goal of this study is to quantify surgeon performance and biometric data to understand how modifiable behaviors can maximize recovery and performance.

DETAILED DESCRIPTION:
Participants will be asked to wear a biometric sensor for six months. The biometric sensor, namely, 'The Whoop strap' collects heart rate and heart rate variability data.

Other data gathered will be in the form of surveys and comments from subjects on wellness, burnout, modifiable activities including sleep, nutrition, exercise and mindfulness, and surgical performance as well as video and audio recordings during a simulated surgical task.

Surveys will be individually numbered and a master list of subject number and video, audio, and sensor ID will be kept in a separate location. This practice will enable us to better understand survey feedback by reviewing relevant videos, images, and sensor recordings. Images and data associated with a subject will be labeled with the subject number only.

ELIGIBILITY:
Inclusion Criteria:

* Study participants will include trainee and attending surgeons

Exclusion Criteria:

* Exclusion criteria will be anyone who is not full-time clinically active as a surgical trainee or attending

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Surgical trainees and attendings at Stanford Health Care
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Surgeon Recovery | 6-12 months
  A daily Recovery score from 0-100% (0-33% is poor recovery, 34-66% is medium recovery, 67-100% is good recovery) is calculated using the WHOOP algorithm which takes resting heart rate, heart rate variability, and sleep metrics into account.

SECONDARY OUTCOMES:
Clinical Strain | 6-12 months
  Strain scores are calculated using the WHOOP algorithm which uses heart rate, activity, and duration of activity. The Clinical Strain will refer to the Strain calculated by the WHOOP strap that occurs during clinical activities including overnight call and operative cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Health Care, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No